CLINICAL TRIAL: NCT03303547
Title: Concordance of Imaging and Pathology Diagnosis of Extranodal Tumour Deposits
Acronym: COMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Pelican Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCUMAS: 23HH8158
Record Dates: First submitted 2017-09-13; First posted 2017-10-06 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Adenocarcinoma of the Rectum
Keywords: MRI; Tissue; Imaging; Pathology; Rectal; Cancer
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI-Pathology N1c matching group (Experimental): MRI mapping will be used to guide pathologists to sample areas of the mesorectum where tumour deposits are likely to be present.
  Interventions: Diagnostic Test: MRI mapping to guide pathological sampling of extranodal tumour deposits

INTERVENTIONS:
Diagnostic Test: MRI mapping to guide pathological sampling of extranodal tumour deposits — Radiologist to mark areas where extranodal disease is identified on MRI. The pathologist will use this to take additional samples for analysis. This will allow better pathological staging and will affect treatment decisions for patients.

SUMMARY:
Any patient with a suspected primary adenocarcinoma of the colon, sigmoid or rectum undergoing surgery are eligible. The date of surgery must be known prior to registration. This trial aims to determine if image mapping techniques can improve the concordance between imaging and pathology detection of tumour deposits. Lymph nodes and tumour deposits will be identified on pre-operative scans and mapped by radiologists then shared with pathologists prior to processing the resected specimen. Patients will be managed at their local hospital with standard follow-up. Patients will be followed up for 5 years.

DETAILED DESCRIPTION:
A prospective interventional multi-centre study, COMET aims to prove the accuracy of imaging diagnosis of extranodal tumour deposits (TD) and their adverse effect on prognosis of colorectal cancers. The proposed intervention will be additional radiological and pathological assessment and the reporting of supplementary diagnostic information which would not otherwise have been available. This may affect treatment according to local MDT protocols and also affect the provision of prognostic information to patients in subsequent discussions.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected primary adenocarcinoma of the colon, sigmoid or rectum (proven by biopsy taken as part of routine clinical practice, patients to be withdrawn if not subsequently adenocarcinoma on pathology).
2. Amenable to surgical resection.
3. Disease spread assessed on imaging
4. Patients having primary surgery and those undergoing neoadjuvant treatment will be included.
5. All must have had baseline staging scans and those undergoing neoadjuvant therapy must also have had a post-treatment scan.
6. Patients aged 16 years and over

Exclusion Criteria:

1. Patients with recurrent tumours
2. Synchronous tumours
3. Under the age of 16 years
4. Unable to give informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-10-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether the prevalence of TD on pathology is found to be higher if imaging mapping is used. | Up to 2 years
  Comparison of the proportion of patients with TD on imaging with proportion of patients with TD on histopathology defined as 'nodules without definite features of lymph node architecture'

SECONDARY OUTCOMES:
To determine whether lesions classified as TD on Imaging correspond to the pathological diagnosis of TD. | Up to 2 years
  Correspondence of nodules identified as tumour deposits on imaging and nodules identified as tumour deposits on the corresponding pathology slice
To determine the effect of Imaging and pathological diagnosis of TD on disease free survival (at one, three and five years), overall survival (at one, three and five years) and time to local recurrence. | 1, 3 and 5 years
  Survival and recurrence outcomes according to Imaging and histopathology TD status
To investigate features of the primary tumour compared with tumour deposits | Up to 2 years and up to 5 years follow up
  Comparison of immunohistochemical and morphological features of tumour
To investigate features of the primary tumour compared with lymph nodes | Up to 2 years and up to 5 years follow up
  Comparison of immunohistochemical and morphological features of tumour
To objectively record the features seen which help distinguish a LN from an TD and attempt to refine and clarify the definitions used in pathology. | Up to 2 years
  Comparison of histopathological known features in patients with MR defined TD vs lymph nodes e.g. capsule, peripheral lymphocyte ring, vessel wall, "lone arteriole sign"
To objectively record the features seen which help distinguish a LN from an TD | Up to 2 years
  Comparison of histopathological known features in patients with MR defined TD vs lymph nodes e.g. capsule, peripheral lymphocyte ring, vessel wall, "lone arteriole sign"
To assess inter-observer agreement between the local pathologist and the central reviewing pathologist. | Up to 2 years0
  Overall comparison of professional agreement between specialists on TD status at recruiting site vs central review - description of location and number of tumour deposits
To assess inter-observer agreement between the local radiologist and central reviewing radiologist. | Up to 2 years
  Overall comparison of professional agreement between specialists on TD status at recruiting site vs central review - description of location and number of tumour deposits

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, MD, Principal Investigator — Imperial College London
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lord AC, Moran B, Abulafi M, Rasheed S, Nagtegaal ID, Terlizzo M, Brown G. Can extranodal tumour deposits be diagnosed on MRI? Protocol for a multicentre clinical trial (the COMET trial). BMJ Open. 2020 Oct 7;10(10):e033395. doi: 10.1136/bmjopen-2019-033395. PMID 33033006